CLINICAL TRIAL: NCT01576926
Title: Evolution of Swallowing in Patients Undergoing Lateral Pharyngoplasty With Preservation Stylopharyngeal Muscle
Status: Completed | Type: Observational
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Principal Investigator, Jayson mesti, evolution of swallowing in patients undergoing lateral pharyngoplasty, Hospital do Servidor Publico Estadual
Other Study IDs: 116/08
Record Dates: First submitted 2012-04-09; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea, obstructive; Deglutition Disorders
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Deglutition Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- surgery: patients with obstructive sleep apnea

SUMMARY:
Evolution of swallowing in patients undergoing lateral pharyngoplasty with preservation stylopharyngeal muscle.

DETAILED DESCRIPTION:
refer patients to the side pharyngoplasty with total preservation of stylopharyngeal muscle and evaluate the total recovery time of swallowing, making a daily assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients with obstructive sleep apnea with surgical indication

Exclusion Criteria:

* patients with obstructive sleep apnea without surgical indication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with obstructive sleep apnea, indicating the lateral pharyngeal
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evolution of swallowing in patients undergoing lateral pharyngoplasty with preservation stylopharyngeal muscle | assess progress daily until the end of swallowing dysphagia during 30 days
  refer patients with oas to the side faringolastia with total preservation stylopharyngeal muscle and evaluate recovery time of swallowing during 30 days.

SECONDARY OUTCOMES:
Evolution of swallowing in patients undergoing lateral pharyngoplasty with preservation stylopharyngeal muscle | assess progress daily until the end of swallowing dysphagia during 30 days
  refer patients with oas to the side faringolastia with total preservation styleopharingeal muscle and evaluate the total recovery time of swallowing, making a daily assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jayson Mesti, medical, Principal Investigator — Hopital Do Servidor Público Estadual
Locations (1):
- Hospital Do Servidor Publico Estadual, São Paulo, São Paulo, Brazil